CLINICAL TRIAL: NCT06886802
Title: Multicentric Case Series of Uniportal Endoscopic Posterior Cervical Decompression for Cervical Spinal Stenosis
Acronym: DEC-SCM
Status: Not yet recruiting | Type: Observational
Sponsor: TecSalud Investigación Clínica (Other)
Collaborators: Tecnologico de Monterrey (Other); Centro Medico Nacional Siglo XXI IMSS (Other); Hospital Ángeles Tijuana (Unknown); TecSalud (Unknown); Hospital Zambrano Hellion TecSalud, Mexico (Unknown)
Responsible Party: Sponsor
Other Study IDs: DEC-SCM
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Spinal Stenosis Cervical
Keywords: Cervical Spinal Stenosis; ► Minimally Invasive Surgical Procedures; ► Endoscopic Spine Surgery; ► Spinal Degenerative Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical Spinal Stenosis Cases: Patients diagnosed with cervical spinal stenosis who exhibit persistent neurological deficits and pain despite receiving at least three months of conservative treatment. All participants have elected to undergo Posterior Uniportal Endoscopic Cervical Decompression. They are being prospectively followed to evaluate improvements in neurological function and reductions in pain-related disability, as well as to document perioperative outcomes including surgical time, blood loss, hospital stay, and complications.
  Interventions: Procedure: Posterior Uniportal Endoscopic Cervical Decompression

INTERVENTIONS:
Procedure: Posterior Uniportal Endoscopic Cervical Decompression — Posterior Uniportal Endoscopic Cervical Decompression

SUMMARY:
Cervical spinal stenosis is a condition that can cause pain, sensory disturbances, and motor deficits due to the compression of neural structures in the cervical spine. While conservative treatments such as physical therapy and pain management can help some patients, others with persistent neurological deficits may require surgical intervention. Traditional surgical approaches, including anterior decompression and posterior open surgery, have proven effective but carry risks such as vascular or nerve injuries and postoperative pain.

This study evaluates a minimally invasive surgical approach called Posterior Uniportal Endoscopic Cervical Decompression as an alternative to traditional methods for patients with cervical spinal stenosis. The main objective is to assess changes in neurological deficits and disability related to cervical pain following this procedure. The study will also document hospitalization duration, surgical time, blood loss, and the incidence of postoperative complications.

This multicenter, prospective case series will recruit 50 patients from three medical centers in Mexico. Participants must have symptomatic cervical spinal stenosis that persists despite at least three months of conservative treatment. Eligible patients will undergo Posterior Uniportal Endoscopic Cervical Decompression, a technique that allows precise nerve decompression through a small incision, minimizing damage to surrounding tissues. Standardized clinical assessment tools, including the modified Japanese Orthopaedic Association (mJOA) scale, Neck Disability Index (NDI), and Visual Analog Scale (VAS) for pain, will be used to evaluate outcomes at multiple time points over 12 months.

By comparing patients' preoperative and postoperative evaluations, the study aims to determine whether Posterior Uniportal Endoscopic Cervical Decompression effectively improves neurological function and reduces disability while maintaining a favorable safety profile. Findings from this study could support the adoption of minimally invasive endoscopic techniques as a viable option for treating cervical spinal stenosis, potentially leading to faster recovery times and reduced surgical complications compared to traditional methods.

DETAILED DESCRIPTION:
Cervical spinal stenosis is a condition characterized by the narrowing of the cervical spinal canal, leading to compression of the neural structures. This can cause chronic pain, sensory disturbances, and motor deficits, significantly impairing the quality of life. While conservative management, including physical therapy, analgesics, and steroid injections, can provide symptomatic relief for some patients, others with persistent neurological deficits may require surgical intervention. Traditional surgical techniques, such as anterior cervical decompression and fusion or posterior open decompression, have been effective but carry risks such as vascular injury, neurological complications, and postoperative pain.

This study investigates the use of Posterior Uniportal Endoscopic Cervical Decompression, a minimally invasive surgical approach that offers targeted decompression through a single small incision while minimizing tissue disruption. The primary objective of the study is to evaluate changes in neurological deficits and disability related to cervical pain following this procedure. Secondary objectives include assessing the duration of hospitalization, surgical time, blood loss, and the incidence of postoperative complications.

This multicenter, prospective case series will recruit 50 patients diagnosed with cervical spinal stenosis at three medical institutions in Mexico. The study will be conducted over a period of 24 months, with an initial 12-month patient recruitment phase, followed by postoperative follow-up assessments at predetermined time intervals up to one year.

Participants will undergo Posterior Uniportal Endoscopic Cervical Decompression, a technique designed to preserve spinal mobility while reducing compression on the nerve roots. The procedure will be performed under general anesthesia with continuous neurophysiological monitoring, including somatosensory evoked potentials, motor evoked potentials, and continuous electromyography. Using a working-channel endoscope, surgeons will perform foraminotomies or laminotomies to remove compressive elements such as osteophytes, hypertrophic ligaments, or herniated disc material. The technique is aimed at achieving decompression with minimal disruption to the surrounding soft tissues.

Patients must meet specific inclusion criteria, including an age range of 18 to 75 years, confirmed diagnosis of cervical spinal stenosis (Kang classification grade I-III), and the presence of neurological symptoms unresponsive to at least three months of conservative management. Exclusion criteria include prior cervical surgery at the affected level, active infections, systemic inflammatory diseases, vertebral instability, congenital spinal malformations, and contraindications for general anesthesia.

Patient outcomes will be systematically evaluated using validated clinical assessment tools, including:

* Modified Japanese Orthopaedic Association (mJOA) Scale - to assess neurological function.
* Neck Disability Index (NDI) - to measure the impact of cervical pain on daily activities.
* Visual Analog Scale (VAS) for pain - to quantify cervical and upper limb pain intensity.
* EQ-5D-5L health-related quality of life questionnaire - to evaluate overall well-being.
* Modified MacNab Criteria - to determine patient satisfaction with surgical outcomes.

Descriptive statistical methods will be used to analyze demographic and clinical characteristics of the study population. Changes in primary and secondary outcomes will be evaluated using paired t-tests for continuous variables and Chi-square tests for categorical variables. The impact of the procedure on neurological function and pain relief will be assessed through longitudinal comparisons between baseline and follow-up assessments at 1, 3, 6, and 12 months postoperatively. The incidence of complications will be categorized using the Clavien-Dindo classification, and the Comprehensive Complication Index will be used to quantify cumulative morbidity.

This study complies with the Declaration of Helsinki, the International Council for Harmonisation Good Clinical Practice (ICH-GCP) guidelines, and national regulatory requirements. All participants will provide written informed consent before enrollment, and patient confidentiality will be maintained through data pseudonymization. The study has been approved by the Ethics Committees of the participating institutions.

The expected impact of this study is to generate clinical evidence supporting Posterior Uniportal Endoscopic Cervical Decompression as a safe and effective alternative to traditional surgical approaches for cervical spinal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent to participate in the study.
* Patients with cervical canal stenosis grade I-III according to the Kang scale.
* Radicular or myelopathic symptoms.
* Having undergone complete conservative management, including physical therapy and analgesia, for at least 3 months.
* Patients who have opted for posterior uniportal endoscopic cervical decompression for cervical canal stenosis.

Exclusion Criteria:

* Inability to read or write.
* Prior cervical surgeries at the levels to be treated.
* Infectious symptoms or concomitant rheumatologic diseases.
* Criteria of cervical vertebral instability.
* Congenital spinal malformations.
* Disc herniation at the same cervical level to be operated on.
* Medullary hyperintensity on T2-weighted magnetic resonance imaging in the level(s) to be treated.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: • Patients with cervical spinal stenosis who continue to experience symptoms despite receiving complete conservative management for at least 3 months and who have chosen to undergo posterior uniportal endoscopic cervical decompression will be recruited consecutively. Recruitment will take place at the following healthcare centers:
  * Centro Médico Zambrano-Hellion, TecSalud (San Pedro Garza García, N.L.) and Clínica Cuauhtémoc y Famosa (Monterrey, N.L.) Patients will be recruited by Dr. Mario Benvenutti Regato, a neurosurgery specialist with over 7 years of experience performing endoscopic spine surgery.
  * Centro Médico Nacional Siglo XXI (Mexico City) Patients will be recruited by Dr. Félix Domínguez Cortinas, a neurosurgery specialist with over 10 years of experience performing endoscopic spine surgery.
  * Hospital Ángeles Tijuana (Tijuana, B.C.) Patients will be recruited by Dr. Alfonso García Chávez, a specialist in traumatology and orthopedics with over 10 years of experience perfor
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Cervical Disability (Neck Disability Index) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure assesses disability related to cervical pain using the Neck Disability Index (NDI), a validated instrument scored from 0 (no disability) to 100 (maximum disability). It quantifies the impact of cervical pain on daily activities and overall function. Changes in NDI scores over time will reflect the effectiveness of the surgical intervention in reducing pain-related disability.
Change in Neurological Function (Modified Japanese Orthopaedic Association Score) | Baseline; 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure evaluates neurological function using the Modified Japanese Orthopaedic Association (mJOA) scale. The mJOA score, which ranges from 0 (severe neurological deficits) to 18 (normal neurological function), assesses motor function, sensory deficits, and gait. Improvements in the mJOA score following surgery will be used as an indicator of enhanced neurological status.

SECONDARY OUTCOMES:
Duration of Hospitalization | Measured during the index hospitalization.
  This metric records the total number of days from patient admission until discharge following the surgical procedure. It serves as an indicator of the immediate postoperative recovery and overall efficiency of the surgical intervention.
Duration of Surgery | Recorded intraoperatively.
  This outcome measures the surgical time, defined as the period from the initial incision to the final closure of the surgical site. It reflects procedural efficiency and may indirectly indicate the technical ease or complexity of the procedure.
Intraoperative Blood Loss | Assessed during the surgical procedure.
  This measure quantifies the volume of blood lost during the surgical procedure, as collected via standard suction devices and measured in milliliters. It is an important indicator of surgical safety and efficiency.
Rate of Perioperative Complications | Assessed 7 days, 1 month, 3 months, 6 months, and 12 months postoperatively.
  This measure records the incidence and severity of complications occurring during the perioperative period. Complications will be categorized according to the Clavien-Dindo classification and summarized using the Comprehensive Complication Index, providing a quantitative assessment of overall surgical morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Benvenutti Regato, MD, Principal Investigator — TecSalud
Locations (1):
- Hospital Zambrano Hellion, TecSalud, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye ZY, Kong WJ, Xin ZJ, Fu Q, Ao J, Cao GR, Cai YQ, Liao WB. Clinical Observation of Posterior Percutaneous Full-Endoscopic Cervical Foraminotomy as a Treatment for Osseous Foraminal Stenosis. World Neurosurg. 2017 Oct;106:945-952. doi: 10.1016/j.wneu.2017.07.085. Epub 2017 Jul 21. PMID 28739520
- [Background] Lv J, Mei J, Feng X, Tian X, Sun L. Clinical efficacy and safety of posterior minimally invasive surgery in cervical spondylosis: a systematic review. J Orthop Surg Res. 2022 Aug 13;17(1):389. doi: 10.1186/s13018-022-03274-3. PMID 35964065
- [Background] Metzger RL. Evidence-based diagnosis and treatment of cervical spine disorders. Nurse Pract. 2019 Aug;44(8):30-37. doi: 10.1097/01.NPR.0000574648.67659.09. PMID 31268958